CLINICAL TRIAL: NCT06872008
Title: Effect Of Hand Massage Applied To Elderly Stayıng In Nursing Homes On Sleep Quality and Anxiety Level: Randomized Controlled Trial
Brief Title: Hand Massage Applied To Elderly Stayıng In Nursing Homes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Amasya University (Other)
Responsible Party: Principal Investigator, Tuğba, Master Student, Amasya University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: AUSBFTSARI001
Record Dates: First submitted 2024-11-26; First posted 2025-03-12 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Sleep Quality; Anxiety Level
Keywords: HAND MASSAGE; SLEEP QUALITY; ANXIETY LEVEL; NURSING HOME; RANDOMIZED CONTROLLED STUDY; ELDERLY
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Participant Group (Experimental): Hand Massage
  Interventions: Behavioral: Hand Massage
- Control Group (No Intervention): No Massage

INTERVENTIONS:
Behavioral: Hand Massage — Hand massage to elderly people Hand massage application consists of five basic classical massages including efflorage, petrissage, friction, tapotman and vibration.
  It is a massage that includes manipulation and is performed with western technique.
  The researcher will collaborate with the institution's physiotherapist throughout the application. Hand massage in the literature Although there is no standard duration for how long the massage should be applied, studies have shown that the massage is applied for an average of 5-10 times, and in this study the massage application time was It was determined as 10 minutes in total, 5 minutes for each hand. Hand massage with baby oil will be performed 3 times a week for 4 weeks, for a total of 12 sessions.
  Arms: Participant Group

SUMMARY:
Hand massage; behavioral and reduce psychological symptoms, enable individuals to calm down and relax, and provide individual and care It is applied to contribute to communication between donors, to ensure reliability and ease of application, to improve the quality of life and to reduce symptoms such as sleep problems, fatigue, pain, stress, anxiety and depression that the individual frequently experiences.

This study will be carried out to determine the effect of hand massage on the sleep quality and anxiety level of elderly people living in nursing homes.

The number of samples of the research G-Power 3.1.9.7 program was used in the calculation. In the analysis, the average scores of the Pittsburgh Sleep Quality Scale were used and 58 individuals (29 experimental, 29 control) were required.

In the research, it was aimed to assign 30 people to each group, taking into account the high power of the test and the losses.

Hand massage in the literature Although there is no standard duration for how long to apply, studies have shown that the massage is applied for an average of 5-10 times, and in this study, the massage application time was It was determined as 10 minutes in total, 5 minutes for each hand. Hand massage with baby oil will be performed 3 times a week for 4 weeks, for a total of 12 sessions.

Research data, Diagnostic Information Form, Pittsburgh Sleep Quality Index (PSQI), Trait Anxiety Scale It will be collected using (STAI-TX). The data obtained from the research were analyzed in the Statistical Package for Social Science (SPSS) 21 statistical program.

will be done. Variables covering the descriptive characteristics of individuals with chronic diseases are expressed in numbers and percentages.

will be done. Whether the data has a normal distribution will be determined by the Shapiro-Wilk test and parametric and/or non-parametric tests will be used depending on the results obtained. Statistical significance value will be accepted as p<05.

DETAILED DESCRIPTION:
Hand massage application consists of five basic classical massages including efflorage, petrissage, friction, tapotman and vibration.

It is a massage that includes manipulation and is performed with western technique. Hand massage; behavioral and psychological symptoms, to enable individuals to calm down and relax, to contribute to communication between individuals and caregivers, to ensure ease of application, to improve quality of life, and to reduce symptoms such as sleep problems, fatigue, pain, stress, anxiety and depression that the individual frequently experiences. is implemented. Easily learned Its important advantages are that it is applicable, non-invasive, does not require position changes and does not cause privacy violations.

ELIGIBILITY:
Inclusion Criteria:

* Being suitable for participation in the study according to the institution's psychosocial report
* Being a nursing home resident and being 60 years of age or older
* Not having been diagnosed with Alzheimer's or dementia
* Being able to speak and understand Turkish
* Not having problems with sensory perception and communication skills
* Not having any problems with applying hand massage
* Giving consent to participate in the study.

Exclusion Criteria:

* Having a cognitive problem
* Hand and nail deformities with thrombus, phlebitis, ecchymosis, hematoma, impaired skin integrity to be,
* Using antidepressant, hypnotic, benzodiazepine and narcotic derivative drugs that affect sleep quality.

Criteria for Discontinuation from Follow-up:

* Wanting to leave after the research has started.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2024-11-18 (Actual); Primary Completion 2024-12-20 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
Pittsburgh Sleep Quality Index | Baseline and week 4
  The Pittsburgh Sleep Quality Index (PSQI) is a 19-item self-report measure that evaluates sleep quality and disturbance over the past month.
  is the scale. It consists of 24 questions, 19 questions are self-report questions, 5 questions are questions to be answered by the spouse or roommate. The 18 scored questions of the scale consist of 7 components. Subjective Sleep Quality, Sleep Latency,Sleep Duration, Habitual Sleep Efficiency, Sleep Disturbance,Sleeping Drug Use and Daytime Dysfunction. Each A component is evaluated on a scale of 0-3 points. The total score of the 7 components gives the scale total score. Total score varies between 0-21. Your total score is less than 5being large indicates "poor sleep quality"
STAI-TX Anxiety Scale | Baseline and week 4
  The transformed expressions in the Trait Anxiety Inventory constitute items 21, 26, 27, 30, 33, 36 and 39. After having the total weights of direct and uttered expressions separately, subtracting the reverse expressions in terms of total weight from the total weight score obtained for direct expressions. A clearly determined and unchanging value is added to this number. The last value obtained is the person's anxiety. The Trait Anxiety Scale (SCSS) indicates that the person shows a persistent level of anxiety about life in general. Scores range from 20 (low anxiety) to 80 (high anxiety)

CONTACTS AND LOCATIONS:
Overall Officials: Tuğba Sarı, MSc, Principal Investigator — Amasya University
Locations (1):
- Amasya University, Amasya, Turkey (Türkiye)